CLINICAL TRIAL: NCT05615285
Title: Personalised Exercise Rehabilitation for Cancer Survivorship
Acronym: PERCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Irish Cancer Society (Other); National Cancer Control Programme, Ireland (Unknown); Trinity St James's Cancer Institute, Dublin, Ireland (Unknown); Royal College of Surgeons, Ireland (Other); Technological University Dublin, Ireland (Unknown); La Trobe University, Melbourne, Australia (Unknown); Wellcome Trust (Other)
Responsible Party: Principal Investigator, Emer Guinan, Assistant Professor, University of Dublin, Trinity College
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PERCS
Record Dates: First submitted 2022-10-21; First posted 2022-11-14 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Cancer
Keywords: Cancer rehabilitation; Exercise; Triage
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: A feasibility and implementation study of the PERCS triage and referral system. Participants are triaged into one of three groups, but the outcomes of the groups will not be compared from an intervention perspective. The system will be evaluated as a whole.
Masking Description: Implementation study designed to operate closely to clinical practice: no masking appropriate or required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PERCS Triage and Referral System — Participants will undergo an assessment of physical function and psychosocial wellbeing. Researchers will apply a triage algorithm, based on findings of assessment. Participants will be referred to one of three exercise-based rehabilitation pathways which will best meet their rehabilitation needs. Participants will be re-assessed after 12 weeks. System will be evaluated using RE-AIM framework.

SUMMARY:
There is strong evidence that exercise can help improve physical and mental wellbeing after treatment for cancer. However, at present, people with cancer in Ireland are not given the opportunity to have an individual assessment of their physical and psychological wellbeing as part of standard care and are not routinely prescribed exercise-based rehabilitation.

The researchers will run and evaluate a system to i. assess physical and psychological wellbeing of people who have completed cancer treatment, ii. apply a rehabilitation triage system, based on findings of the assessment, iii. refer participants to one of three rehabilitation pathways, as per outcome of the triage process.

Rehabilitation pathways are as follows:

1. Participants who are currently active and have no cancer-specific impairments will receive advice from the physiotherapist on maintaining their current levels of activity.
2. Participants who are not active and have no cancer-specific impairments will be referred to a suitable community-based exercise programme. This programme must contain both resistance and aerobic training and should have some level of supervision from a fitness professional.
3. Participants who are not active and have ongoing cancer-specific impairments will be referred to an oncology specialist physiotherapist, funded through this work, at St James's Hospital for assessment and treatment.

All participants will be encouraged to visit www.cancerrehabilitation.ie for information through out the study. Participants will be reassessed 12 weeks after the initial assessment.

The implementation of this system will be evaluated using the RE-AIM framework.

DETAILED DESCRIPTION:
Background During and following treatment for cancer, people can experience negative side-effects of treatment, including loss of fitness, weakness, fatigue and psychological issues such as depression and anxiety. There is strong evidence that exercise can help improve these symptoms. The impact of the COVID-19 pandemic means that many people who had cancer treatment since March 2020 may need additional support to achieve optimum physical and psychological wellbeing. At present, people with cancer in Ireland are not given the opportunity to have an individual assessment of their physical and psychological wellbeing as part of standard care and are not routinely prescribed exercise-based rehabilitation.

Aim To run and evaluate an exercise-based rehabilitation triage and assessment clinic for people who had cancer treatment since the beginning of the COVID-19 pandemic.

Study Design:

Patients who were diagnosed with cancer in St James Hospital since March 2020 will be invited to participate in the study. Participants will attend an appointment with a physiotherapist, who will assess their physical and mental wellbeing. On the basis of the assessment findings, participants will be assigned to one of three categories, which will determine their ongoing rehabilitation plan. The three categories are as follows:

1. Participants who are currently active and have no cancer-specific impairments will receive advice from the physiotherapist on maintaining their current levels of activity.
2. Participants who are not active and have no cancer-specific impairments will be referred to a suitable community-based exercise programme. This programme must contain both resistance and aerobic training and should have some level of supervision from a fitness professional.
3. Participants who are not active and have ongoing cancer-specific impairments will be referred to an oncology specialist physiotherapist, funded through this work, at St James's Hospital for assessment and treatment.

All participants will also be advised to visit a website designed by the PERCS research group through a co-design process with patient representatives (www.cancerrehabilitation.ie.) Participants will receive a follow-up phone call one week after the first assessment and will then be re-assessed 12 weeks after the first assessment. A further follow-up phone call will be conducted, if the PERCS research team feel it is needed.

The assessment and triage clinic will be assessed using a framework for evaluating intervention; this will look at how the intervention was implemented and how it will best operate in future practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible to participate if they:

  1. Were diagnosed with cancer at St James's Hospital since March 2020
  2. Have completed adjuvant chemotherapy and/or radiotherapy
  3. Are at least 6 weeks post-surgery
  4. Do not show signs of recurrent or metastatic disease at the time of enrolment
  5. Are over the age of 18 years

     Exclusion Criteria:

     Anyone who is unable to provide informed consent Any person with known or signs or symptoms suggestive of cardiovascular, metabolic or renal disease will require medical clearance from a physiotherapist or medical professional prior to participation, based on criteria outlined in the Safety Reference Guide to support the safe delivery of exercise services to people with cancer by Santa Mina et al. (2018). Preparticipation screening will be completed in accordance with the American College of Sports Medicine Preparticipation health screening recommendations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
RE-AIM Framework | Data reported by 12 months
  Evaluation of system Reach, Effectiveness, Adoption, Implementation, Maintenance
Percentage of patients on Prehabilitation list which are eligible for the study | Data reported by 12 months
  Referral - Eligible referral rate from prehabilitation group
The percentage of referrals to the study from clinical team which are eligible for the study | Data reported by 12 months
  Referral - Eligible referral rate from clinical teams
Percentage of people enrolled in study who have received both recruitment letter and phone call | Data reported by 12 months
  Enrolment rate
Percentage of people attending scheduled assessments at i. T0 and ii. T1 | Data reported by 12 months
  Assessment completion rate
Percentage of people who attended assessment who proceed to attend level 2 or level 3 referral service | Data reported by 12 months
  Attrition rate - referrals
Percentage of people who attended T0 assessment that attend T1 assessment | Data reported by 12 months
  Attrition rate - assessments
i. Time from assessment to referral being sent ii. Percentage of referral accepted at initial site iii. Time from referral sent to initial appointment | Data reported by 12 months
  Referral outcome - time frame and acceptance
i. Percentage of people triaged to each level (1, 2 or 3) ii. Percentage triaged to another level after initial triage and why | Data reported by 12 months
  Triage results
Number and nature of adverse events occurring in assessment process | Data reported by 12 months
  Adverse events
Information related to feasibility gathered from semi-structured interviews with participants | Data reported by 12 months
  Qualitative feasibility

SECONDARY OUTCOMES:
International Physical Activity Questionnaire | T0 assessment, T1 (+12 weeks from T0 assessment); data reported by 12 months
  Physical activity levels assessment Health Behaviour and Stages of Change Questionnaire Self-Efficacy for Exercise Scale
Health Behaviour and Stages of Change Questionnaire | T0 assessment, T1 (+12 weeks from T0 assessment); data reported by 12 months
  Readiness to change assessment Health Behaviour and Stages of Change Questionnaire Self-Efficacy for Exercise Scale
Self-efficacy for exercise scale | T0 assessment, T1 (+12 weeks from T0 assessment); data reported by 12 months
  Physical activity self efficacy assessment Health Behaviour and Stages of Change Questionnaire Self-Efficacy for Exercise Scale
Patient specific funcational scale | T0 assessment, T1 (+12 weeks from T0 assessment); data reported by 12 months
  Self-reported function. Scale from 0 - 10, higher score indicates higher perceived ability to do task
Timed Up and Go | T0 assessment, T1 (+12 weeks from T0 assessment); data reported by 12 months
  Falls Risk
Hand grip strength | T0 assessment, T1 (+12 weeks from T0 assessment); data reported by 12 months
  Muscle strength
30 second Sit-to-Stand | T0 assessment, T1 (+12 weeks from T0 assessment); data reported by 12 months
  Funcational lower body strength
Six minute walk test | T0 assessment, T1 (+12 weeks from T0 assessment); data reported by 12 months
  aerobic capacity &endurance
Height | T0 assessment, T1 (+12 weeks from T0 assessment); data reported by 12 months
  Anthropometrics
Weight | T0 assessment, T1 (+12 weeks from T0 assessment); data reported by 12 months
  Anthropometrics
Waist Circumference | T0 assessment, T1 (+12 weeks from T0 assessment); data reported by 12 months
  Anthropometrics
Mid-arm Circumference | T0 assessment, T1 (+12 weeks from T0 assessment); data reported by 12 months
  Anthropometrics
Mini Nutritional Assessment | T0 assessment, T1 (+12 weeks from T0 assessment); data reported by 12 months
  Nutritional
EOCG-PS | T0 assessment, T1 (+12 weeks from T0 assessment); data reported by 12 months
  Performance status
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC- QLQ-C30) | T0 assessment, T1 (+12 weeks from T0 assessment); data reported by 12 months
  Quality of life
Multidimensional Fatigue Inventory (MFI-20) | T0 assessment, T1 (+12 weeks from T0 assessment); data reported by 12 months
  Fatigue
Hospital Anxiety and Depression Scale (HADS) | T0 assessment, T1 (+12 weeks from T0 assessment); data reported by 12 months
  Anxiety & depression; Scale from 0 - 21, higher score indicates higher levels of anxiety and/or depression.
Sociodemographic details | T0 assessment; data reported by 12 months
Medical history | T0 assessment; data reported by 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Facility, St James's Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brennan L, Kennedy M, Grehan S, Connolly H, Sheill G, Donohoe CL, Guinan E. Patient experiences of participating in a cancer rehabilitation triage and referral system in the Irish healthcare system. J Cancer Surviv. 2025 Mar 27. doi: 10.1007/s11764-025-01785-6. Online ahead of print. PMID 40146479
- [Derived] Brennan L, Sheill G, Collier S, Browne P, Donohoe C, Guinan E. Personalised exercise rehabilitation in cancer survivorship: Findings from a triage and referral feasibility study. J Cancer Surviv. 2024 Nov 12. doi: 10.1007/s11764-024-01684-2. Online ahead of print. PMID 39528780
- [Derived] Brennan L, Sheill G, Collier S, Browne P, Donohoe CL, O'Neill L, Hussey J, Guinan EM. Personalised exercise rehabilitation in cancer survivorship: the percs triage and referral system study protocol. BMC Cancer. 2024 Apr 23;24(1):517. doi: 10.1186/s12885-024-12266-x. PMID 38654198